

# Device Protocol for CLY935-C018 / NCT05056987 Title: Clinical Assessment of Two Daily Wear Reusable Soft Silicone Hydrogel Contact Lenses

Protocol Number: CLY935-C018

Clinical Investigation

Type:

Test Product:

TOTAL30 contact lens (lehfilcon A)

Sponsor Name and Alcon Research, LLC, and its affiliates ("Alcon")

Interventional

Address: 6201 South Freeway

Fort Worth, Texas 76134-2099

Property of Alcon Confidential

May not be used, divulged, published, or otherwise disclosed without the consent of Alcon

Document ID: V-CLN-0002831

Page 2 of 65

Status: Approved, Version: 3.0 Approved Date: 02 Dec 2021

#### Investigator Agreement:

- I have read the clinical study described herein, recognize its confidentiality, and agree to conduct the described trial in compliance with Good Clinical Practices; applicable international and national regulations, laws, guidelines, and standards; the conditions of approval imposed by the reviewing IRB or regulatory authority; and in accordance with the ethical medical research principles outlined in the Declaration of Helsinki.
- I will supervise all testing of the device involving human subjects and ensure that the requirements relating to obtaining informed consent and IRB review and approval are met in accordance with applicable local and governmental regulations.
- I have read and understand the appropriate use of the investigational product(s) as described in the protocol, current investigator's brochure, product information, or other sources provided by the sponsor.
- I understand the potential risks and side effects of the investigational product(s).
- I agree to maintain adequate and accurate records in accordance with government regulations and to make those records available for inspection.
- I agree to comply with all other requirements regarding the obligations of clinical investigators and all other pertinent requirements of the sponsor and government agencies.
- I agree to ensure that all associates, colleagues, and employees assisting in the conduct of the study are informed of their obligations in meeting the above commitments.

| | Have you ever been disqualified as an investigator by any Regulatory Authority? | | | | |
|---|---|---|---|---|---|
| | □ No | □Yes | | | |
| | Have you | ever been i | involved in a stud | dy or other research that was | terminated? |
| | □ No | □Yes | | | |
| | If yes, ple | ease explain | here: | | |
| Pr | incipal inv | estigator: | | | |
| | | | Signature | | Date |
| | ame and prosition: | ofessional | | | |
| Αc | ddress: | | | | |
| Ph | one Numb | er: | | | |
| | Off-hours Emergency<br>Phone Number: | | | | |

# **Table of Contents**

| De | vice Prote | ocol for CLY935-C018 | 1 |
|---|---|---|---|
| Ta | ble of Co | ntents | 3 |
| Lis | st of Table | es | 5 |
| Lis | st of Figu | res | 6 |
| 1 | GLOSS | ARY OF TERMS | 7 |
| 2 | LIST OF | F ACRONYMS AND ABBREVIATIONS | 13 |
| 3 | PROTO | COL SUMMARY | 15 |
| 4 | PROTO | COL AMENDMENTS | 22 |
| 5 | INTROI | DUCTION | 22 |
| | 5.1 | Rationale and Background | |
| | 5.2 | Purpose of the Study | |
| | 5.3 | Risks and Benefits | |
| 6 | STUDY | OBJECTIVES | 24 |
| | 6.1 | Primary Objective(s) | 24 |
| | 6.2 | Secondary Objective(s) | 24 |
| | 6.4 | Safety Objective(s) | |
| 7 | INVEST | ΓΙGATIONAL PLAN | 26 |
| | 7.1 | Study Design | 26 |
| | 7.2 | Rationale for Study Design. | 27 |
| | | 7.2.1 Purpose and Timing of Interim Analyses and Resulting Design Adaptations | 20 |
| | 7.3 | Rationale for Duration of Treatment/Follow-Up | |
| | 7.4 | Rationale for Choice of Comparator Product | |
| | 7.5 | Data Monitoring Committee | 28 |
| 8 | STUDY | POPULATION | 28 |
| | 8.1 | Inclusion Criteria | 28 |
| | 8.2 | Exclusion Criteria | 29 |
| | 8.3 | Rescreening of Subjects | 30 |
| 9 | TREATI | MENTS ADMINISTERED | 31 |

| | 9.1 | Investigational Product(s) | 31 |
|---|---|---|---|
| | 9.2 | Other Medical Device or Medication Specified for Use During the Study | <sup>,</sup> 35 |
| | 9.3 | Treatment Assignment / Randomization | 35 |
| | 9.4 | Treatment masking | 36 |
| | 9.5 | Accountability Procedures | 37 |
| | 9.6 | Changes to concomitant medications, treatments/ procedures | 38 |
| 10 5 | STUDY | PROCEDURES AND ASSESSMENTS | |
| | 10.1 | Informed Consent and Screening | 39 |
| | 10.2 | Description of Study Procedures and Assessments | |
| | | 10.2.1 Demographics | |
| | | 10.2.2 Medical History and Concomitant Medications | |
| | | 10.2.3 Investigational Product compliance | |
| | | 10.2.4 Adverse Event Collection: Safety Assessment | 40 |
| | | 10.2.5 Slit Lamp Biomicroscopy: Safety Assessment | 40 |
| | | 10.2.6 Device Deficiencies: Safety Assessment | |
| | | 10.2.7 Additional Study Assessments | |
| | 10.3 | Unscheduled Visits | 41 |
| | 10.4 | Discontinued Subjects | 41 |
| | | 10.4.1 Screen Failures | 41 |
| | | 10.4.2 Discontinuations | 42 |
| | | 10.4.3 Schedule of Procedures and Assessments for Subjects Discontinued from Investigational Product | 42 |
| | 10.5 | Clinical Study Termination | 42 |
| | | 10.5.1 Follow-up of subjects after study participation has ended | 43 |
| 11 / | ADVER | SE EVENTS AND DEVICE DEFICIENCIES | 43 |
| | 11.1 | General Information | 43 |
| | 11.2 | Monitoring for Adverse Events | 45 |
| | 11.3 | Procedures for Recording and Reporting | 46 |
| | 11.4 | Return product analysis, if applicable | 48 |
| | 11.5 | Unmasking of the Study Treatment | 48 |
| | 11.6 | Follow-Up of Subjects with Adverse Events | 49 |
| | 11.7 | Pregnancy in the Clinical Study | |
| 12 | ANALY | SIS PLAN | |
| | 12.1 | Subject Evaluability | 50 |

| 12.2 | Analysis Sets. | .50 |
|------------|----------------------------------------------------------|-----|
| | 12.2.1 Safety Analysis Set | .50 |
| 12.3 | Demographic and Baseline Characteristics | .50 |
| 12.4 | Effectiveness Analyses | .50 |
| | 12.4.1 Analysis of Primary Effectiveness Endpoint(s) | |
| | 12.4.1.1 Statistical Hypotheses | .50 |
| 12.5 | Handling of Missing Data | .52 |
| 12.6 | Safety Analyses | .52 |
| 12.7 | Sample Size Justification | |
| 13 DATA HA | ANDLING AND ADMINISTRATIVE REQUIREMENTS | .53 |
| 13.1 | Subject Confidentiality | .53 |
| 13.2 | Completion of Source Documents and Case Report Forms | .53 |
| 13.3 | Data Review and Clarifications | .54 |
| 13.4 | Sponsor and Monitoring Responsibilities | .54 |
| 13.5 | Regulatory Documentation and Records Retention | .55 |
| 13.6 | Quality Assurance and Quality Control | .55 |
| 14 ETHICS | | .55 |
| | List of Tables | |
| Table 2–1 | List of Acronyms and Abbreviations Used in This Protocol | .13 |
| Table 3–1 | Schedule of Study Procedures and Assessments | .20 |
| Table 6–1 | Primary Objective(s) | .24 |

| Document ID:<br>V-CLN-000283 | Status: Approved, Version: 3.0 Approved Date: 02 Dec 2021 | Page 6 of 65 |
|---|---|---|
| Table 6–3 | Safety Objective(s) | 25 |
| Table 9–1 | Test Product | 31 |
| Table 9–2 | Comparator Product | 33 |
| Table 9–3 | Unmasked Sponsor Members Associated with the Study | 36 |
| | List of Figures | |
| Figure 11-1 | Categorization of All Adverse Events | 43 |
| Figure 11-2 | Categorization of All Serious Adverse Events | 44 |

# 1 GLOSSARY OF TERMS

| Names of test product(s) | Throughout this document, test product(s) will be referred to as TOTAL30® soft contact lenses (TOTAL30) |
|---|---|
| Name of Comparator<br>Product(s) | Throughout this document, comparator product(s) will be referred to as ACUVUE OASYS® with HYDRACLEAR® PLUS contact lenses (AOHP) |
| Adverse Device Effect (ADE) | Adverse event related to the use of an investigational medical device (investigational product) or control product. Note: This definition includes adverse events resulting from insufficient or inadequate instructions for use, deployment, implantation, installation, or operation; any malfunction; and use error or intentional misuse of the investigational medical device (investigational product) or control product. |
| Adverse Event (AE) | Untoward medical occurrence, unintended disease or injury, or untoward clinical signs (including abnormal laboratory findings) in subjects, users or other persons, whether or not related to the investigational medical device (investigational product). |
| | Note: This definition includes events related to the investigational medical device, comparator, or the procedures involved. For users or other persons, this definition is restricted to events related to the use of investigational medical devices (investigational product) or control product. |
| | Requirements for reporting Adverse Events in the study can be found in Section 11. |

| Clinical Investigation Plan (CIP) | The document(s) stating the rationale, objectives, design, and prespecified analysis, methodology, organization, monitoring, conduct, and record-keeping of the clinical investigation. Note: The protocol and other documents referenced in the protocol (for example, the Statistical Analysis Plan, the Manual of Procedures, the Deviations and Evaluability Plan, and the Protocol Monitoring Plan) comprise the CIP. |
|---|---|
| Clinical Investigation Report (CIR) / Clinical Study Report | The document describing the design, execution, statistical analysis, and results of a clinical investigation. The Clinical Investigation Report is synonymous with the Clinical Study Report. |
| Device Deficiency | Inadequacy of a medical device with respect to its identity, quality, durability, reliability, usability, safety, or performance. Note: This definition includes malfunctions, use errors, and inadequacy in the information supplied by the manufacturer including labelling. Requirements for reporting Device Deficiencies in the study can be found in Section 11. |
| Enrolled Subject | Any subject who signs an informed consent form for participation in the study. |
| Point of Enrollment | The time at which, following recruitment and before any clinical investigation-related procedures are undertaken, a subject signs and dates the informed consent form. |
| Interventional Clinical Trial | A pre- or postmarket clinical investigation where the assignment of a subject to a particular medical device is decided in advance by a clinical investigation plan, or diagnostic or monitoring procedures requested in the CIP are in addition to those available as normal clinical practice and burden the subject. |

| Investigational Product | A preventative (vaccine), a therapeutic (drug or biologic), device, diagnostic, or palliative used as a test or comparator product in a clinical trial, including a product with a marketing authorization when used or assembled (formulated or packaged) in a way different from the authorized form, or when used for an unauthorized indication, or when used to gain further information about the authorized form. |
|---|---|
| Malfunction | Failure of an investigational medical device to perform in accordance with its intended purpose when used in accordance with the instructions for use or clinical investigation plan (CIP). |
| Nonserious Adverse Event | Adverse event that does not meet the criteria for a serious adverse event. |
| Product Complaint | Any oral, electronic, or written communication that alleges deficiencies related to the identity (labeling), quality, durability, reliability, safety, effectiveness, or performance of a marketed product, including failure of the product, labeling, or packaging to meet specifications, whether or not the product is related to or caused the alleged deficiency. A complaint may allege that an adverse event or medical device malfunction has occurred. |
| Randomized Subject | Any subject who is assigned a randomized treatment. |
| Serious Adverse Device<br>Effect (SADE) | Adverse device effect that has resulted in any of the consequences characteristic of a serious adverse event. |

# Serious Adverse Event (SAE)

Adverse event that led to any of the following:

- Death.
- A serious deterioration in the health of the subject, users or other persons as defined by one or more of the following:
  - a) a life-threatening illness or injury *Note: Life-threatening means that the individual was* at immediate risk of death from the event as it occurred, i.e., it does not include an event which hypothetically might have caused death had it occurred in a more severe form.
  - b) any potentially sight-threatening event or permanent impairment to a body structure or a body function including chronic diseases.
  - c) inpatient hospitalization or prolonged hospitalization.

Note: Planned hospitalization for a preexisting condition, without serious deterioration in health, is not considered a serious adverse event. In general, hospitalization signifies that the individual remained at the hospital or emergency ward for observation and/or treatment (usually involving an overnight stay) that would not have been appropriate in the physician's office or an outpatient setting. Complications that occur during hospitalization are adverse events. If a complication prolongs hospitalization or fulfills any other serious criteria, the event is serious. When in doubt as to whether "hospitalization" occurred, the event should be considered serious.

- d) a medical or surgical intervention to prevent a) or b).
- e) any indirect harm as a consequence of incorrect diagnostic test results when used within manufacturer's instructions for use.

| | Fetal distress, fetal death, congenital abnormality or birth defect including physical or mental impairment. |
|---|---|
| | Note: Planned hospitalization for a preexisting condition, or a procedure required by the CIP, without serious |
| | deterioration in health, is not considered a serious adverse event. |
| | Refer to Section 11 for additional SAEs. |
| Serious Health Threat | Signal from any adverse event or device deficiency that |
| | indicates an imminent risk of death or a serious deterioration |
| | in the health in subjects, users, or other persons, and that |
| | requires prompt remedial action for other subjects, users, or other persons. |
| | Note: This would include events that are of significant and unexpected nature such that they become alarming as a potential serious health hazard or possibility of multiple deaths occurring at short intervals. |
| Study Start | The start of the study is considered to coincide with the enrollment of the first patient. |
| Study Completion | The completion of the study is considered to coincide with |
| | the database lock or the decision to terminate the trial, whichever is later. |

| Use Error | User action or lack of user action while using the medical |
|---|---|
| | device that leads to a different result than that intended by |
| | the manufacturer or expected by the user. |
| | Note: |
| | a) Use error includes the inability of the user to complete a task. |
| | b) Use errors can result from a mismatch between the characteristics of the user, user interface, task, or use environment. |
| | c) Users might be aware or unaware that a use error has occurred. |
| | d) An unexpected physiological response of the patient |
| | is not by itself considered a use error. |
| | e) A malfunction of a medical device that causes an |
| | unexpected result is not considered a use error." |

# 2 LIST OF ACRONYMS AND ABBREVIATIONS

Table 2–1 List of Acronyms and Abbreviations Used in This Protocol

| Abbreviation | Definition |
|-----------------|------------------------------------------------------|
| ADE | Adverse device effect |
| AE | Adverse event |
| AOHP soft | ACUVUE OASYS with HYDRACLEAR PLUS (AOHP) (senofilcon |
| contact lens or | (A) |
| AOHP | , |
| AOS | Advanced Ophthalmic Systems |
| BCVA | Best corrected visual acuity |
| CE | Conformitè Europëenne |
| CFR | Code of Federal Regulations |
| CIP | Clinical Investigation Plan |
| CIR | Clinical Investigation Report |
| COL | Clinical operations lead |
| CRF | Case report form |
| CSM | Clinical site manager |
| CTT | Clinical trial team |
| D | Diopter(s) |
| eCRF | Electronic case report form |
| EDC | Electronic data capture |
| FDA | US Food and Drug Administration |
| GCP | Good Clinical Practice |
| GPCMS | Global Product Complaint Management System |
| hr | Hour |
| IB | Investigator's brochure |
| ICF | Informed consent form |
| IEC | Independent ethics committee |
| IFU | Instructions for use |
| IP | Investigational product |
| IRB | Institutional review board |
| ISO | International Organization for Standardization |
| logMAR | Logarithm of the minimum angle of resolution |
| mm | Millimeter |
| MOP | Manual of procedures |
| N/A | Not applicable |
| OD | Right eye |
| OS | Left eye |
| SADE | Serious adverse device effect |
| SAE | Serious adverse event |
| SD | Standard deviation |

Document ID: V-CLN-0002831

| Abbreviation | Definition |
|--------------------------------------------|------------------------------|
| SLE | Slit lamp examination |
| SOP | Standard operating procedure |
| TOTAL30 soft<br>contact lens or<br>TOTAL30 | TOTAL30 soft contact lenses |
| UK | United Kingdom |
| US / USA | United States of America |
| USV | Unscheduled visit |
| VA | Visual acuity |

# **3 PROTOCOL SUMMARY**

| Investigational | Device |
|---|---|
| product type | |
| T · | |
| Study type | Interventional |
| Investigational | Test Product: TOTAL30 soft contact lenses (TOTAL30) |
| products | |
| | Comparator Product: ACUVUE OASYS with HYDRACLEAR |
| | PLUS soft contact lenses (AOHP) |
| Purpose and | The overall objective of this clinical study is to describe the |
| Scientific Rationale | clinical performance of the TOTAL30 soft contact lens compared |
| for the Study | to the AOHP soft contact lens in a daily wear modality. |
| V | |
| Objective(s) | The <b>primary objective</b> is to evaluate visual acuity of the |
| | TOTAL30 soft contact lens and the AOHP soft contact lens. |
| Endpoint(s) | Primary Effectiveness |
| | Distance VA (logMAR) with study lenses |

Safety Adverse events Biomicroscopy findings Device deficiencies Assessment(s) Effectiveness Distance VA (logMAR) with study lenses



| Subject population | Volunteer subjects aged ≥ 18 years who are any habitual spherical soft contact lens wearers, have at least 3 months of contact lens wearing experience, and who would be willing to wear the study lenses for at least 5 days per week and at least 8 hours per day. Pregnant and breastfeeding women are excluded for this study. Planned number of subjects enrolled/consented: ~36 Planned number of completed subjects: 32 |
|---|---|
| Sites and Locations | Planned number of clinical sites: 1 |
| | Planned locations (initial list of locations, which may change during start up or conduct according to study needs): UK |
| Key inclusion criteria (See Section 8.1 for a complete list of inclusion criteria) | <ul> <li>Current wearers of any commercial spherical soft contact lenses with at least 3 months wearing experience, who would be willing to wear the study lenses for a minimum wearing time of 5 days per week and 8 hours per day.</li> <li>Able to wear contact lenses within a range of sphere power from -1.00 D to -6.00 D (0.25 D steps) and subject willing and able to wear the study lenses for the full duration of the study.</li> <li>Willing to NOT use rewetting/lubricating drops at any time during the study.</li> </ul> |
| Key exclusion criteria (See Section 8.2 for a complete list of exclusion criteria) | <ul> <li>Participation of the subject in a clinical trial within the previous 14 days or currently enrolled in any clinical trial.</li> <li>Habitual AOHP contact lens wearers (in the past 3 months)</li> <li>Monovision wear during the study.</li> </ul> |
| Data analysis and sample size justification | Planned Analysis To address the primary objective, descriptive statistics (number of observations, mean, standard deviation, median, minimum, maximum) for visual acuity, collected for each eye, on the logMAR scale will be provided. No inferential testing will be conducted. |

| | Sample Size Justification |
|---|---|
| | Given the feasibility nature of this study, sample size calculation is not relevant. |
| Associated materials | AOSEPT PLUS with HydraGlyde Cleaning & Disinfecting |
| | Solution will be used for daily cleaning and disinfection. |
| | Lubrication/rewetting drops will not be permitted during this study. |

Table 3-1 Schedule of Study Procedures and Assessments

| | | | LENS | S PAIR 1 | | LENS PAIR 2 | | |
|---|---|---|---|---|---|---|---|---|
| Procedure/ Assessment | Pre-screening | ì | Visit 1<br>Screen/Baseline/<br>Dispense Pair 1 | Dispense Pair 2 | 1 | Visit 3<br>Follow-up Pair<br>2 <sup>\$</sup> /Exit | Early | USV |
| Trocedure/ Assessment | SC | | Visit V | Window $^{\Omega}$ | | Visit Window Ω | Exit | CSV |
| | | | Day 1 | <b>AOHP</b> = [Day 14<br>(-3/+7 days)]<br><b>TOTAL30</b> = [Day<br>28 (-3/+7 days)] | | AOHP = [Day 14<br>(-3/+7 days)]<br>TOTAL30 = [Day<br>28 (-3/+7 days)] | | |
| Pre-Screening Consent | X | | | | | | | |
| Informed Consent | | | X | | | | | |
| Demographics | | | X | | | | | |
| Medical History* | | | X | X | | X | X | X |
| Pregnancy Form* | | | | (X) | | (X) | (X) | X |
| Concomitant Medications* | | | X | X | | X | X | X |
| Inclusion/Exclusion | | | X | | | | | |
| Habitual (lens brand, lens power*,<br>lens care) | | | X | | | | | |
| Keratometry readings (OD, OS) | | | X | | | | | |
| Manifest refraction* | | | X | (X) | | (X) | (X) | (X) |
| BCVA* (OD, OS, logMAR distance with manifest refraction) | | | X | (X) | | (X) | (X) | (X) |
| Biomicroscopy | | | X | X | | X | X | (X) |
| Randomization | | | X | | | | | |
| VA w/ study lenses, (OD, OS, logMAR distance) | | | X<br>(optimization and<br>baseline<br>measurements for<br>both study lens<br>types) | X<br>(lens pair 1) | | X<br>(lens pair 2) | X | X |
| Slit-lamp photo/video of study lenses* | | | (X) | (X) | | (X) | (X) | (X) |
| Dispense (provide) study lenses | | | X | X | | | | (X) |

| Procedure/ Assessment | | | LENS PAIR 1 | | | LENS PAIR 2 | | |
|---|---|---|---|---|---|---|---|---|
| | | 1 | Visit 1<br>Screen/Baseline/<br>Dispense Pair 1 | Visit 2<br>Follow-up Pair 1 <sup>\$</sup> /<br>Dispense Pair 2 | ì | Visit 3<br>Follow-up Pair<br>2 <sup>\$</sup> /Exit | Early<br>Exit | USV |
| Troccourc/ Assessment | -sc | | Visit Window <sup>Ω</sup> | | | Visit Window <sup>Ω</sup> | | |
| | Pre-screening | | Day 1 | AOHP = [Day 14<br>(-3/+7 days)]<br>TOTAL30 = [Day<br>28 (-3/+7 days)] | | AOHP = [Day 14<br>(-3/+7 days)]<br>TOTAL30 = [Day<br>28 (-3/+7 days)] | | |
| Subjective VAS questionnaire | | | X<br>(baseline<br>measurements for<br>both study lens | X<br>(lens pair 1) | | X<br>(lens pair 2) | X | (X) |

| _ | | | | | |
|---------------------|-----|-----|---|---|-----|
| AEs | X | X | X | X | X |
| Device deficiencies | X | X | X | X | X |
| Exit Form | (X) | (X) | X | X | (X) |

<sup>(</sup>X) Assessment performed as necessary, eg, decrease of VA by 2 lines or more with investigational product (IP)  $USV = Unscheduled\ Visit$ 

<sup>\*</sup> Source only

Subjects are required to wear the study lenses at least 6 hrs on the day of follow-up visits prior to the visit. Follow-up visit time to be within ±2 hours of baseline visit time.

 $<sup>^{\</sup>Omega}$ Visit 2 and 3 visit window and exposure period is dependent on the randomized treatment sequence. AOHP exposure period is to be 14 days (-3/+7 days) and TOTAL30 exposure period is to be 28 days (-3/+7 days)

#### 4 PROTOCOL AMENDMENTS

Modification of the protocol is prohibited without prior written agreement in the form of a protocol amendment. All amendments must be created by the study sponsor and must be approved by the IRB/IEC and global and regional Health Authorities, as applicable, prior to implementation except when required to mitigate immediate safety risks or when the changes involve only logistical or administrative revisions.

Amendments may necessitate that the informed consent and other study-related material be revised. If the consent form is revised, all subjects currently enrolled in the study must sign the approved, revised informed consent (re-consent), as required by the IRB/IEC.

#### 5 INTRODUCTION

### 5.1 Rationale and Background

Daily wear contact lenses are worn during waking hours, often for a full day and then removed for cleaning and disinfection prior to reinsertion the following day. Frequent replacement daily wear contact lenses are replaced according to the product package insert/IFU provided by the contact lens manufacturer.

New silicone hydrogel materials continue to be developed, possessing unique material properties and superior oxygen transmissibility over contact lenses made with conventional hydrogel materials. A new lens, known as the TOTAL30 contact lens, has been developed in an effort to maintain sustained performance by providing an inherently wettable core material with a water gradient surface. The new silicone hydrogel lens has been designed to provide favorable performance for daily wear with 1-month replacement.

In this clinical study, the clinical performance of the TOTAL30 contact lens will be assessed and the TOTAL30 contact lens will be compared to the AOHP contact lens in a crossover design, both to be worn in a daily wear modality.

# 5.2 Purpose of the Study

The purpose of this study is to assess the clinical performance of the TOTAL30 contact lens compared to AOHP. The primary endpoint was selected to address the primary objective of the study. Procedures for measurement of these endpoints were selected based on common practice for these assessments and some novel assessment techniques. The design of this study is justified based upon preclinical and clinical testing, as described within the IFU.

Document ID: V-CLN-0002831

Status: Approved, Version: 3.0 Approved Date: 02 Dec 2021

AOHP contact lenses were chosen as the comparator product because both of these lenses have a frequent replacement schedule.

| At the end of the study, a clinical study report will be prepared in ecordance with applicable regulatory requirements and standards. |
|---|
| Alcon reserves the right of prior review of any publication or presentation of information |
| elated to the study. |

#### 5.3 Risks and Benefits

The clinical investigation process risks are managed through appropriate training and monitoring according to the protocol-specific monitoring plan. Investigational device risks, including risks associated with use of device and methods and procedures for application of device, are defined in the investigator's brochure and/or product labeling and are managed through review of safety assessments outlined in this protocol.

Contact lenses may offer improved peripheral vision and the convenience of not wearing spectacles. Material properties and design characteristics of the study contact lenses are features consistent with successful contact lens wear.

TOTAL30 and AOHP contact lenses are commercially available for daily wear use under a frequent replacement wear modality; further details on any known potential risks and benefits can be found in the IFU.

A summary of the known potential risks and benefits associated with the TOTAL30 and AOHP contact lenses can be found in the IFU. There may also be unknown risks to use of the TOTAL30 contact lens. Any risk to subjects in this clinical study will be minimized by compliance with the eligibility criteria and study procedures, clinical oversight and monitoring, and through close supervision by a licensed clinician during exposure to the study lenses. The site personnel will educate subjects on proper hygiene and lens handling, as

well as compliance with the use of contact lenses and lens care according to the protocol. Subjects should be instructed not to wear contact lenses while sleeping or swimming.

The site personnel will also advise the subjects to remove contact lenses and return for prompt follow-up of symptoms, such as ocular discomfort, foreign body sensation, excessive tearing, vision changes, or hyperemia.



#### **6 STUDY OBJECTIVES**

# 6.1 Primary Objective(s)

Table 6–1 Primary Objective(s)

| Objective(s) | Endpoint(s) |
|---|---|
| To evaluate visual acuity of the TOTAL30 | Distance VA with study lenses (OD, OS; |
| soft contact lens and the AOHP soft contact | logMAR) |
| lens. | |

# **6.2** Secondary Objective(s)

Not Applicable.



# 6.4 Safety Objective(s)

Table 6–3 Safety Objective(s)

| Objective(s) | Endpoint(s) |
|---|---|
| Describe the safety profile of the study | • AEs |
| products | <ul> <li>Biomicroscopy findings</li> </ul> |
| | <ul> <li>Device deficiencies</li> </ul> |

#### 7 INVESTIGATIONAL PLAN

#### 7.1 Study Design

This is a prospective, randomized, bilateral crossover, controlled, subject-masked, daily wear clinical study to be conducted at a single site. Eligible habitual soft contact lens wearers will be randomized to 1 of the 2 crossover sequences. Subjects will be masked. A designated study staff member will prepare the contact lenses for dispensing.

Subjects will be expected to participate in a pre-screening and attend 3 office visits: Screen/Baseline/Dispense Lens Pair 1, Follow-up Lens Pair 1/Dispense Lens Pair 2, Follow-up Lens Pair 2/Exit. AOHP will be worn for  $\sim$ 14 days and TOTAL30 will be worn for  $\sim$ 28 days. The total expected duration of participation for each subject is approximately 1.5 months. Subjects will be randomized to wear the assigned product sequence in both eyes, either the test TOTAL30 contact lenses as Pair 1, followed by the comparator AOHP contact lenses as Pair 2, or vice versa. All study contact lenses will be prescribed according to subject's prescription and can be optimized per study lens type, however test and comparator lenses should be dispensed within  $\pm$ 0.25 D of each other.

Subjects will be expected to wear their study contact lens in a daily wear modality for at least 5 days per week 8 hours a day, over a 14 day (AOHP) or 28 day period (TOTAL30). AOSEPT PLUS with HydraGlyde Cleaning & Disinfecting Solution will be used for daily cleaning and disinfection.

On the day of Visits 2 and 3, subjects will be asked to wear the study lenses at least 6 hours and prior to their study visit. Follow-up visit time to be within  $\pm 2$  hours of baseline visit time.



# 7.2 Rationale for Study Design

study.

This study design is justified based upon an evaluation of the results of relevant preclinical and clinical testing, as described within the IFU.

The crossover design will ensure that the same subject is exposed to both the test and comparator lens materials

The study will include only those subjects who are current wearers of spherical soft contact lenses in both eyes with at least 3 months wearing experience, with a minimum wearing time of 5 days per week and 8 hours per day.

Furthermore, the subjects will not be permitted to use lubrication/rewetting drops during the duration of the study as this may confound the primary effectiveness endpoint. The study will exclude any habitual AOHP contact lens wearers in the past 3 months prior to consent in order to reduce potential bias of wearers to their habitual contact lenses. The study will also

exclude subjects who wish to wear their contact lenses in monovision modality during the

# 7.2.1 Purpose and Timing of Interim Analyses and Resulting Design Adaptations

An interim analysis will not be performed.

## 7.3 Rationale for Duration of Treatment/Follow-Up

Subjects will wear the test and comparator products bilaterally for approximately 28 and 14 days, depending on the lens being dispensed. Subjects will remain masked to the lens type. The primary variable will be assessed on Day 1 and at Day 28 for test product and at Day 14 for comparator product.

#### 7.4 Rationale for Choice of Comparator Product

AOHP contact lenses were chosen as the comparator product because these lenses have the same wear modality and similar replacement schedule.

# 7.5 Data Monitoring Committee

Not applicable.

#### 8 STUDY POPULATION

The study population consists of male and female subjects (aged 18 or over) who are current wearers of spherical soft contact lenses in both eyes with a least 3 months wearing experience, with a minimum wearing time of 5 days per week and 8 hours per day. Subjects who are habitual AOHP contact lens wearers in the past 3 months will be excluded. It is aimed to enroll (consent) approximately 36 subjects at 1 site in the United Kingdom, with a target of 32 completed subjects

Estimated time needed to recruit subjects for the study is approximately 5 months; however, unanticipated circumstances may shorten or lengthen this time and would not require amendment of this protocol. Eligible study population will be representative of the study products target population.

#### 8.1 Inclusion Criteria

Written informed consent must be obtained before any study specific assessment is performed. Upon signing informed consent, the subject is considered enrolled in the study.

- 1. Subjects must be  $\geq$  18 years of age and have capacity to volunteer.
- 2. Subjects must be able to understand and must sign an informed consent form (ICF) that has been approved by an Institutional Review Board (IRB/IEC).
- 3. Current wearers of any commercial spherical soft contact lenses with at least 3 months wearing experience, who would be willing to wear the study lenses for a minimum wearing time of 5 days per week and 8 hours per day.
- 4. Manifest cylinder  $\leq 0.75$  D in each eye (based on the ocular refraction).
- 5. Able to wear contact lenses within a range of sphere power from -1.00 D to -6.00 D (0.25 D steps) and subject willing and able to wear the study lenses for the full duration of the study.
- 6. Best corrected distance visual acuity better than or equal to 0.10 logMAR in each eye (as determined by manifest refraction at screening).
- 7. Subjects must be willing to stop wearing their habitual contact lenses for the duration of study participation.
- 8. Subjects must be willing to NOT use rewetting/lubricating drops at any time during the study



#### 8.2 Exclusion Criteria

Subjects fulfilling **any** of the following criteria are not eligible for participation in this study.

- 1. Any anterior segment infection, inflammation, or abnormality or disease (including systemic) that contraindicates contact lens wear, as determined by the investigator.
- 2. Any use of systemic or ocular medications for which contact lens wear could be contraindicated, as determined by the investigator.
- 3. History of refractive surgery or plan to have refractive surgery during the study or irregular cornea in either eye.

- 4. Ocular or intraocular surgery (excluding placement of punctal plugs) within the previous 12 months or planned during the study.
- 5. Biomicroscopy findings at screening that are moderate (Grade 3) or higher and/or corneal vascularization that is mild (Grade 2) or higher; presence of corneal infiltrates.
- 6. Current or history of pathologically dry eye in either eye that, in the opinion of the investigator, would preclude contact lens wear.
- 7. Current or history of herpetic keratitis in either eye.
- 8. Eye injury in either eye within twelve weeks immediately prior to enrollment for this trial.
- 10. Any use of topical ocular medications and artificial tear or rewetting drops that would require instillation during the study.
- 11. The investigator, his/her staff, family members of the investigator, family members of the investigator's staff, or individuals living in the households of the aforementioned persons may not participate in the study.
- 12. Participation of the subject in a clinical trial within the previous 14 days or currently enrolled in any clinical trial.
- 13. Monovision wear during the study.
- 14. Habitual AOHP contact lens wearers (in the past 3 months)
- 15. Currently pregnant or breast-feeding.

# 8.3 Rescreening of Subjects

Rescreening of subjects is not allowed in this study.

## 9 TREATMENTS ADMINISTERED

#### 9.1 **Investigational Product(s)**

*Test Product(s):* TOTAL30 soft contact lenses (TOTAL30)

Comparator Product(s) (If

AOHP (senofilcon A) soft contact lenses

applicable):

Table 9–1 **Test Product** 

| Test Product | TOTAL30 soft contact lenses (TOTAL30) |
|---|---|
| Manufacturer | Alcon Laboratories, Inc. 6201 South Freeway Fort Worth, Texas 76134-2099 USA |
| Indication for use and intended purpose in the current study | The intended use of this product is for vision correction. |
| Product description<br>and parameters<br>available for this<br>study | <ul> <li>Material: lehfilcon A</li> <li>Water content: 55%</li> <li>Power range: -1.00 to -6.00 D (0.25 D steps)</li> <li>Base curve (mm): 8.4</li> <li>Diameter (mm): 14.2</li> </ul> |
| Formulation | Silicone hydrogel. For additional details, please refer to the TOTAL30 IFU. |
| Usage | <ul> <li>Wear: <ul> <li>Daily Wear</li> <li>Bilateral</li> <li>Crossover according to randomization</li> </ul> </li> </ul> |

| Number/Amount of product to be provided to the subject | <ul> <li>Replacement period: This is a monthly replacement lens, however lenses will not have a planned replacement in this study.</li> <li>Exposure: At least 8 hours per day, 5 days per week, over a 28 day period.</li> <li>Lens Care: AOSEPT PLUS with HydraGlyde Cleaning &amp; Disinfecting Solution will be used for daily cleaning and disinfection.</li> <li>Additional details can be found in the MOP.</li> <li>Subjects will be dispensed study lenses at Visit 1 and Visit 2. One spare pair of lenses will be provided to the subject.</li> </ul> |
|---|---|
| Packaging description | Blister foil pack |
| Labeling description | <ul> <li>Lens Foil label includes (at a minimum): <ul> <li>lens identifier</li> <li>base curve</li> <li>diameter</li> <li>packing solution</li> <li>power</li> <li>lot number</li> <li>expiration date</li> <li>content statement</li> <li>investigational device statement</li> <li>sponsor information</li> <li>Country of origin</li> </ul> </li> <li>Provided in packages of approximately 72 lenses per power, identified with the following: <ul> <li>a color coded label stating the protocol number</li> <li>material identifier</li> <li>power</li> <li>an investigational use only statement</li> <li>tracking number</li> </ul> </li> </ul> |

| Training and/or | No additional training or experience is required to administer the |
|---|---|
| experience | test product. |
| requirements for | |
| device | |
| Storage conditions | Stored at room temperature. |
| Supply | Alcon will provide a bulk inventory of lenses for the site to use |
| | throughout the trial for fitting and dispense. |
| | Contact lens solution and contact lens case will be provided to the |
| | subject. |

Table 9–2Comparator Product

| Comparator | ACUVUE OASYS with HYDRACLEAR PLUS (AOHP) |
|---|---|
| Product(s) | (senofilcon A) soft contact lenses |
| Manufacturer | Johnson & Johnson |
| Indication for Use | The intended use of this product is for vision correction. |
| Product description | Material: senofilcon A |
| and parameters | • Water content: 38% |
| available for this | • Power range: -1.00 to -6.00 D (0.25 D steps) |
| study | • Base curve (mm): 8.4, 8.8 |
| | • Diameter (mm): 14.0 |
| Formulation | Silicone Hydrogel. For additional details, please refer to the AOHP |
| | IFU. |
| Usage | • Wear: |
| | <ul> <li>Daily Wear</li> </ul> |
| | o Bilateral |
| | <ul> <li>Crossover according to randomization</li> </ul> |
| | • Replacement period: This is a 2 week replacement lens, |
| | however lenses will not have a planned replacement in this |
| | study. |
| | • Exposure: At least 8 hours per day, 5 days per week, over a 14 |
| | day period. |

| Number/Amount of Product to be Provided to the subject | <ul> <li>Lens Care: AOSEPT PLUS with HydraGlyde Cleaning &amp; Disinfecting Solution will be used for daily cleaning and disinfection.</li> <li>Additional details can be found in the MOP.</li> <li>Subjects will be dispensed study lenses at Visit 1 and Visit 2. One spare pair of lenses will be provided to the subject.</li> </ul> |
|---|---|
| Packaging description | Blister foil pack |
| Labeling description | <ul> <li>Lens Foil label includes (at a minimum): <ul> <li>lens identifier</li> <li>base curve</li> <li>diameter</li> <li>packing solution</li> <li>power</li> <li>lot number</li> <li>expiration date</li> <li>content statement</li> <li>investigational device statement</li> <li>sponsor information</li> <li>Country of origin</li> </ul> </li> <li>Provided in packages of approximately 72 lenses per power, identified with the following: <ul> <li>a color coded label stating the protocol number</li> <li>material identifier</li> <li>power</li> <li>an investigational use only statement</li> <li>tracking number</li> </ul> </li> </ul> |
| Training and/or experience requirements for device | No additional training or experience is required to administer the comparator product. |

| Storage conditions | Lenses to be stored at room temperature. |
|---|---|
| Supply | Alcon will provide a bulk inventory of lenses for the site to use throughout the trial for fitting and dispense. Contact lens solution and contact lens case will be provided to the subject. |

More information on the test and comparator products can be found in their individual IFUs.

# 9.2 Other Medical Device or Medication Specified for Use During the Study

During the clinical study, additional contact lens solution is required in conjunction with the treatment:

 AOSEPT PLUS with HydraGlyde Cleaning & Disinfecting Solution will be used for daily cleaning and disinfection.

# 9.3 Treatment Assignment / Randomization

Subjects will be randomized in a 1:1 ratio to receive treatment in crossover sequence of test product then comparator product or comparator product then test product, respectively.



Only after signing the ICF at Visit 1, a subject will be assigned a subject number by the electronic data capture system.

A randomization list will be generated using a validated system that automates the random assignment of treatment arms to randomization numbers in the specified ratio. Subjects will be assigned treatment according to the randomization list uploaded in the randomization system. The randomization list will be generated and maintained by the study sponsor.

At Visit 1, all eligible subjects will be randomized via the EDC/randomization integration system to one of the treatment arms (lens sequences). The investigator's delegate will access the respective system after confirming that the subject meets all the eligibility criteria. A randomization number will be automatically assigned to the subject according to the subject

randomization list but will not be communicated to the site user. The EDC/randomization integration system will inform the site user of the treatment sequence assignment to be dispensed to the subject.

# 9.4 Treatment masking

This study is subject-masked, with subjects randomized to use the TOTAL30 contact lenses and AOHP contact lenses for the duration of the 28 and 14 day treatment period, respectively.




This level of masking will be maintained throughout the conduct of the study. Unmasking will occur only after all planned study data have been validated, and the database locked.

# 9.5 Accountability Procedures

Upon receipt of the IPs, the investigator or delegate must conduct an inventory. During the study, it is recommended that the investigator delegates staff to provide the IPs to the subjects in accordance with their randomization assignment. All members associated with the study at the site should make an attempt to remain masked, except for designated staff who will be dispensing IP and completing IP dispensation and collection records. These records must be made available to the study monitor for the purposes of verifying the accounting of IP supplies. Any discrepancies and/or deficiencies between the observed disposition and the written account must be recorded along with an explanation. All IPs sent to the investigator must be accounted for by study sponsor personnel, and in no case be used in an unauthorized situation.

It is the investigator's responsibility to ensure that:

- All study products are accounted for and not used in any unauthorized manner
- All unused products are available for return to the study sponsor, as directed
- All used lidding foils are available for return to the study sponsor, as directed

Any study lenses associated with a device deficiency or with any product-related adverse
event (i.e., ADE or SADE) are returned to the study sponsor for investigation, unless
otherwise directed by the sponsor. Refer to Section 11 of this protocol for additional
information on the reporting of device deficiencies and AEs and the return of study
products associated with these events.

The investigator is responsible for proper disposition of all unused IPs at the conclusion of the study, according to the instructions provided in the MOP.

# 9.6 Changes to concomitant medications, treatments/ procedures

After the subject is enrolled into the study, the investigator must instruct the subject to notify the study site about:

- Any new medications
- Alterations in dose or dose schedules for current medications
- Any medical procedure or hospitalization that occurred or is planned
- Any nondrug therapies (including physical therapy and blood transfusions)

The investigator must document this information in the subject's case history source documents.

#### 10 STUDY PROCEDURES AND ASSESSMENTS

| Visit # | Visit Type | Visit Day | Visit Window |
|---|---|---|---|
| Visit 1 | Screen/Baseline/Dispense Pair 1 | Day 1 | N/A |
| Visit 2 | Follow-up Pair 1 (Dispense Pair 2)<br>AOHP: Day 14<br>TOTAL30: Day 28 | Day 14<br>Day 28 | Days 11-21<br>Days 25-35 |
| Visit 3 | Follow-up Pair 2/Exit<br>AOHP: Day 14<br>TOTAL30: Day 28 | Day 14<br>Day 28 | Days 11-21<br>Days 25-35 |

Unscheduled Visits and Early Termination Visits are allowed, if necessary.

Study lenses will be provided to the subjects to take home for daily wear during the course of the trial.

Study randomization will occur at Visit 1 with assigned lenses provided to take home at Visit 1 and Visit 2. Study contact lens fitting will occur at Visit 1 for both study lenses. If a subject cannot be successfully fit (either study lens) according to the study lens fitting guides as determined by the investigator, they will be required to exit from the study.

Lubrication/rewetting drops will not be permitted during this study.

#### 10.1 Informed Consent and Screening

The investigator or delegate must explain the purpose and nature of the study, and have the subject read, sign, and date the IRB/IEC-approved informed consent document. The subject must sign the ICF BEFORE any study-specific procedures or assessments can be performed, including study-specific screening procedures. Additionally, have the individual obtaining consent from the subject and a witness, if applicable, sign and date the informed consent document.

The investigator or delegate must provide a copy of the signed document to the subject and place the original signed document in the subject's chart, or provide documentation as required by local regulations.

# 10.2 Description of Study Procedures and Assessments

Study-specific procedures and assessments described here may include standard of care; other standard of care procedures performed in the clinical management of the subject are not excluded.

Detailed descriptions of assessments and procedures are provided in the MOP. All study procedures and assessments are to be performed according to the table of procedures (Table 3-1). The investigator is responsible for ensuring responsibilities for all procedures and assessments are delegated to appropriately qualified site personnel.

# 10.2.1 Demographics

Obtain demographic information including age, race, and sex.

#### **10.2.2 Medical History and Concomitant Medications**

Ocular and non-ocular medical history and concomitant medications will be collected at Visit 1 (and at other visits as needed, i.e., due to AE) and documented in the source documents. All relevant medical conditions, including currently active conditions, diagnosed chronic conditions, and conditions resolved within the past year will be documented. Habitual lens information and medications taken within 30 days prior to Visit 1 will be recorded in the source documentation. Include herbal therapies, vitamins, and all over-the-counter as well as prescription medications. Throughout the subject's participation, obtain information on any changes in medical health and/or the use of concomitant medications and record in subject source documents.

# **10.2.3** Investigational Product compliance

Review subject compliance with the IP usage and adjunct product usage and collect all used and unused study IPs and other products that were dispensed.

# 10.2.4 Adverse Event Collection: Safety Assessment

Assess and record any adverse events that are observed or reported, including those associated with changes in concomitant medication dosing since the previous visit in the subject source documents. See Section 11 for further details regarding AE collection and reporting.

# 10.2.5 Slit Lamp Biomicroscopy: Safety Assessment

SLE of the cornea, iris/anterior chamber, and lens must be performed in both eyes before instillation of any diagnostic eye drops.

# 10.2.6 Device Deficiencies: Safety Assessment

Assess and record any Device Deficiencies that are reported or observed since the previous visit. Requirements for reporting device deficiencies in the study can be found in Section 11. Device deficiencies on comparator lenses should be reported per the manufacturer's guidelines.

# **10.2.7** Additional Study Assessments

Additional effectiveness assessments will be conducted throughout the course of the study. Refer to the MOP and Table 3-1 for details on each of these assessments.

#### 10.3 Unscheduled Visits

If a subject visit occurs between any regularly scheduled visit and the visit is conducted by study personnel, this visit must be documented as an Unscheduled Visit. If the subject seeks medical attention outside the clinic (for example, at an Emergency Room) or at the clinic but is seen by nonstudy personnel, the investigator is to capture adverse event-related information on the Adverse Event form upon becoming aware.

During all unscheduled visits, the investigator must conduct the following procedures:

- Collect Adverse Event information
- Collect device deficiency information
- Record changes in medical condition (including pregnancy) or concomitant medication
- VA with study lenses

The investigator may perform additional procedures for proper diagnosis and treatment of the subject according to Table 3-1 or at their discretion. The investigator must document this information in the subject's case history source documents and in the eCRF, where applicable.

If during an Unscheduled Visit the subject is discontinuing the IP or discontinuing from the study, the investigator must conduct Exit procedures according to Table 3-1 Schedule of Study Procedures and Assessments and Section 10.4.3, as possible.

# 10.4 Discontinued Subjects

#### 10.4.1 Screen Failures

Subjects who were excluded from the study after signing the informed consent and prior to randomization to product/dispense of study product.

The investigator must document the reason for screen failure in the subject's case history source documents and in EDC.

Subject numbers must not be re-used.

#### 10.4.2 Discontinuations

Discontinued subjects are individuals who voluntarily withdraw or are withdrawn from the study by the investigator after signing informed consent.

Subject numbers of discontinued subjects must not be re-used (i.e., subject replacement is not allowed).

Subjects may discontinue from study or study treatment at any time for any reason. Subjects may also be discontinued from study treatment at any time if, in the opinion of the investigator, continued treatment poses a risk to their health.

For subjects discontinuing from the study, the investigator must complete all Exit procedures according to Table 3-1 Schedule of Study Procedures and Assessments if the subject is willing and able, and if in the opinion of the investigator it is safe for the subject to do so.

The investigator must document the reason for study or treatment discontinuation in the subject's case history source documents.

To ensure the safety of all subjects who discontinue early, investigators must assess each subject and, if necessary, advise them of any therapies and/or medical procedures that may be needed to maintain their health.

# 10.4.3 Schedule of Procedures and Assessments for Subjects Discontinued from Investigational Product

Other than screen failures, if a subject discontinues from the study, the subject should undergo an Early Exit Visit. Refer to Table 3-1.

# 10.5 Clinical Study Termination

The study sponsor reserves the right to suspend or close the investigational site or suspend or terminate the study in its entirety at any time.

If the clinical study is prematurely terminated or suspended by the study sponsor:

- The study sponsor must:
  - o Immediately notify the investigator(s) and subsequently provide instructions for study termination.
  - Inform the investigator and the regulatory authorities of the termination/suspension and the reason(s) for the termination/suspension.

#### • The investigator must:

- Promptly notify the IRB/IEC of the termination or suspension and of the reasons.
- Provide subjects with recommendations for poststudy treatment options as needed.

The investigator may terminate the site's participation in the study for reasonable cause.

Breaking of the masked treatment codes will be done after locking the database.

# 10.5.1 Follow-up of subjects after study participation has ended

Following this study, the subject will return to their eye care professional for their routine eye care.

#### 11 ADVERSE EVENTS AND DEVICE DEFICIENCIES

#### 11.1 General Information

An AE is any untoward medical occurrence, unintended disease or injury, or untoward clinical signs (including abnormal laboratory findings) in subjects, users, or other persons, whether or not related to the investigational medical device (test product). Refer to the Glossary of Terms and figures below for categories of AEs and SAEs.

Figure 11-1 Categorization of All Adverse Events



Figure 11-2 Categorization of All Serious Adverse Events



Status: Approved, Version: 3.0

Approved Date: 02 Dec 2021

#### **Specific Events Relevant to this Protocol**

#### Serious Adverse Events

In addition to reporting all AEs (serious and non-serious) meeting the definitions, the investigator must report any occurrence of the following as an SAE:

- An ocular infection including a presumed infectious ulcer with any of the following characteristics:
  - Central or paracentral location
  - o Penetration of Bowman's membrane
  - o Infiltrates > 2 mm diameter
  - o Iritis
  - Increase in intraocular pressure
  - Culture positive for microorganisms
  - Increasing size or severity at subsequent visits
- Any central or paracentral corneal event (such as neovascularization) that results in permanent opacification
- Hypopyon

Document ID: V-CLN-0002831

Status: Approved, Version: 3.0 Approved Date: 02 Dec 2021

- Hyphema
- Neovascularization within the central 6 mm of the cornea
- Permanent vision loss as defined by loss of 2 or more lines of BCVA (i.e., Study Lens Distance VA with Over-Refraction or Manifest Refraction BCVA) from enrollment visit that fails to resolve
- Uveitis (anterior, intermediate, or posterior)
- Corneal abrasion affecting ≥50% of corneal surface area

The above events are based on the categories provided in the ISO 11980 and the US FDA Premarket Notification (510(k)) Guidance Document for Daily Wear Contact Lenses.

#### **Device Deficiencies**

A device deficiency is inadequacy of a medical device with respect to its identity, quality, durability, reliability, safety, or performance. A device deficiency may or may not be associated with patient harm (i.e., ADE or SADE); however, not all ADEs or SADEs are due to a device deficiency. The investigator should determine the applicable category listed in the Device Deficiency eCRF for the identified or suspect device deficiency and report any patient harm separately. Examples of device deficiencies include the following:

- Failure to meet product specifications (e.g., incorrect lens power/diameter/base curve/color)
- Lens/solution cloudy
- Lens surface/edge defect
- Torn lens during handling/in pack
- Packaging deficit (e.g., mislabeled product, tampered seal, leaking bottle/container)
- Suspect product contamination
- Lack of performance

# 11.2 Monitoring for Adverse Events

At each visit, after the subject has had the opportunity to spontaneously mention any problems, the investigator should inquire about AEs by asking the standard questions shown below and report as applicable:

"Have you had any health problems since your last study visit?"

• "Have there been any changes in the medicines you take since your last study visit?"

In addition, changes in any *protocol-specific parameters* evaluated during the study are to be reviewed by the investigator. Any untoward (unfavorable and unintended) change in a *protocol-specific parameter* that is clinically relevant, in the opinion of the investigator, is to be reported as an AE. These clinically relevant changes will be reported regardless of causality.

# 11.3 Procedures for Recording and Reporting

AEs are collected from the time of informed consent. Any pre-existing medical conditions or signs/symptoms present in a subject prior to the start of the study (i.e., before informed consent is signed) are not considered AEs in the study and should be recorded in the Medical History section of the eCRF.

In addition, temporary lens awareness or visual changes during the fitting process are not considered AEs if the investigator assesses that the symptom(s) can reasonably resolve within the anticipated adaptation period.



For each recorded event, the ADEs and SAEs documentation must include: date of occurrence, severity, treatment (if applicable), outcome, and assessments of the seriousness and causality. In addition, the investigator must document all device deficiencies reported or observed with test and comparator products on the Device Deficiency eCRF. The site must submit all available information on ADEs, SAEs, and device deficiencies to the study sponsor immediately as follows:

- All SAEs must be reported immediately (within 24 hours) of the Investigator's or site's awareness.
- ADEs that do not meet seriousness criteria and device deficiencies must be reported within 10 calendar days of the Investigator's or site's awareness.
- A printed copy of the completed Serious Adverse Event and Adverse Device Effect and/or Device Deficiency eCRF must be included with product returns. Additional relevant

information after initial reporting must be entered into the eCRF as soon as the data become available.

- Document any changes to concomitant medications on the source.
- Document all relevant information from Discharge Summary, Autopsy Report,
- Certificate of Death etc., if applicable, in narrative section of the *Serious Adverse Event* and Adverse Device Effect eCRF.

Note: Should the EDC system become non-operational, the site must complete the appropriate paper *Serious Adverse Event and Adverse Device Effect and/or Device Deficiency* Form. The completed form is emailed to the study sponsor at qa.complaints@alcon.com according to the timelines outlined above; however, the reported information must be entered into the EDC system once it becomes operational.

Any AEs and device deficiencies for non-study marketed devices/products (i.e., AOSEPT PLUS with HydraGlyde Cleaning & Disinfecting Solution) will be considered and processed as spontaneous (following the post-market vigilance procedures) and should be communicated to the device's/product's manufacturer as per local requirements.

Study sponsor representatives may be contacted for any protocol related question and their contact information is provided in the Manual of Procedures that accompanies this protocol.

Further, depending upon the nature of the AE or device deficiency being reported, the study sponsor may request copies of applicable portions of the subject's medical records. The investigator must also report all AEs and device deficiencies that could have led to a SADE according to the requirements of regulatory authorities or IRB/IEC.

#### **Intensity and Causality Assessments**

Where appropriate, the investigator must assess the intensity (severity) of the AE based on medical judgment with consideration of any subjective symptom(s), as defined below:

#### Intensity (Severity)

Mild An AE is mild if the subject is aware of but can easily tolerate the sign or symptom.

Moderate An AE is moderate if the sign or symptom results in discomfort significant enough to cause interference with the subject's usual activities.

Severe

An AE is severe if the sign or symptom is incapacitating and results in the subject's inability to work or engage in their usual activities.

For every AE in the study, the investigator must assess the causality (Related or Not Related to the medical device or study procedure). An assessment of causality will also be performed by study sponsor utilizing the same definitions, as shown below:

#### **Causality**

Related

An AE classified as related may be either definitely related or possibly related where a direct cause and effect relationship with the medical device or study procedure has not been demonstrated, but there is a reasonable possibility that the AE was caused by the medical device or study procedure.

Not Related

An AE classified as not related may either be definitely unrelated or simply unlikely to be related (i.e., there are other more likely causes for the AE).

The study sponsor will assess the AEs and may upgrade the investigator's assessment of seriousness and/or causality. The study sponsor will notify the investigator of any AEs that is upgraded from non-serious to serious or from unrelated to related.

# 11.4 Return product analysis, if applicable

Study sponsor representatives and their contact information are provided in the MOP that accompanies this protocol.

Alcon products associated with device deficiencies and/or product related AEs should be returned and must include the Complaint # which will be provided by study sponsor after the case is entered in the study sponsor's Global Product Complaint Management System (GPCMS).

# 11.5 Unmasking of the Study Treatment

Investigators are unmasked in this study. However, the identity of the assigned medical device should not be disclosed to subjects who are masked during the study. The Study Sponsor must be informed of all cases in which unmasking of the subject(s) has occurred and of the circumstances involved. The Study Sponsor should be informed in advance of unmasking when possible, except in the event of a medical emergency. Additionally, the

Study Sponsor may be required to unmask the information in order to fulfill expedited regulatory reporting requirements.

# 11.6 Follow-Up of Subjects with Adverse Events

The investigator is responsible for adequate and safe medical care of subjects during the study and for ensuring that appropriate medical care and relevant follow-up procedures are maintained after the study.

The investigator should provide the study sponsor with any new safety information (which includes new AEs and changes to previously reported AEs) that may affect the safety evaluation of the device. For AEs that are unresolved/ongoing at time of subject exit from study, any additional information received at follow-up should be documented in the eCRFs up to study completion (i.e., database lock).

Any additional data received up to 3 months after subject discontinuation or exit must be documented and available upon the study sponsor's request. All complaints received after this time period will be considered and processed as spontaneous (following the post-market vigilance procedures) and should be communicated to the medical device's manufacturer as per local requirements.

The investigator should also report complaints on non-Alcon products directly to the manufacturer as per the manufacturer's instructions or local regulatory requirements.

# 11.7 Pregnancy in the Clinical Study

Pregnancy is excluded at the time of enrollment for this study. However, if a subject becomes pregnant during study participation, it will be documented on the source. Pregnancy is not reportable as an AE; however, complications may be reportable and will be decided on a case-by-case basis.

#### 12 ANALYSIS PLAN

Continuous variables will be summarized using the number of observations, mean, SD, median, minimum, and maximum. Categorical variables will be summarized with frequencies and percentages from each category.

Any deviations to the analysis plan will be updated during the course of the study as part of a protocol amendment or will be detailed in the clinical study report.

# 12.1 Subject Evaluability

Final subject evaluability must be determined prior to breaking the code for masked treatment (lens) sequence assignment and locking the database, based upon the Deviations and Evaluability Plan.

# 12.2 Analysis Sets

# 12.2.1 Safety Analysis Set

Safety analyses will be conducted using the safety analysis set on a treatment-emergent basis. As such, the safety analysis set will include all subjects/eyes exposed to any study lenses evaluated in this study, \_\_\_\_\_\_\_\_\_. For treatment-emergent safety analyses, subjects/eyes will be categorized under the actual study lenses exposed in the corresponding lens sequence.

# 12.3 Demographic and Baseline Characteristics

Demographic and baseline characteristics will be summarized by lens sequence and overall. Frequencies and percentages will be presented for categorical variables such as sex, age group, and race. Number of observations, mean, SD, median, minimum, and maximum will be presented for continuous variables such as age.

# 12.4 Effectiveness Analyses

This study defines one primary endpoint . The Safety Analysis Set will be used

# 12.4.1 Analysis of Primary Effectiveness Endpoint(s)

The primary objective of this study is to evaluate the VA of the TOTAL30 soft contact lens and the AOHP soft contact lens. The primary endpoint is distance VA with study lenses, collected for each eye in logMAR.

# 12.4.1.1 Statistical Hypotheses

No inferences are to be made on the primary effectiveness endpoint; therefore, no hypotheses are formulated.

# 12.4.1.2 Analysis Methods

Descriptive statistics used for continuous variables will be presented.

# 12.5 Handling of Missing Data

All data obtained in evaluable subjects/eyes will be included in the analysis. No imputation for missing values will be carried out.

# 12.6 Safety Analyses

The safety endpoints are:

- AEs
- Biomicroscopy findings
- Device deficiencies

There are no safety hypotheses planned in this study. The focus of the safety analysis will be a comprehensive descriptive assessment of occurrence of adverse events as well as the other listed parameters.

All AEs occurring from the time a subject signs informed consent to study exit will be accounted for in the reporting. Safety analyses will be conducted using the safety analysis set on a treatment-emergent basis. Descriptive summaries (counts and percentages) for ocular and nonocular AEs will be presented by Medical Dictionary for Regulatory Activities Preferred Terms. AEs leading to study discontinuation, significant non-serious AEs, and SAEs will be identified. Individual subject listings will be provided, as necessary.

Individual subject listings will be provided for AEs that occur after signing informed consent but prior to exposure to IP.

Each biomicroscopy parameter will be tabulated by its grade. For each biomicroscopy parameter, counts and percentages of eyes that experience an increase of  $\geq 2$  grades from baseline (last assessment prior to study lens exposure for each period) to any subsequent visit within the same period will be presented. A supportive listing will be generated which will include all biomicroscopy data from all visits within the same period for those eyes experiencing the increase.

Two listings for device deficiencies, prior to exposure of study contact lenses and treatmentemergent, will be provided. Additionally, each device deficiency category will be tabulated.

No inferential testing will be done for safety analysis.

# 12.7 Sample Size Justification

Given the feasibility nature of this study, sample size calculation is not relevant.

#### 13 DATA HANDLING AND ADMINISTRATIVE REQUIREMENTS

# 13.1 Subject Confidentiality

The investigator must ensure that the subject's identity is kept confidential throughout the course of the study. In particular, the investigator must keep an enrollment log with confidential identifying information that corresponds to the subject numbers and initials of each study participant. The study sponsor may collect a copy of the enrollment log without any identifying subject information.

The study sponsor may share patient-level data collected in this trial with qualified researchers to help facilitate product development or enhancements in research that is not directly related to the study objectives. The Informed Consent explains this to the study subject.

# 13.2 Completion of Source Documents and Case Report Forms

The nature and location of all source documents will be identified to ensure that original data required to complete the CRFs exist and are accessible for verification by the site monitor, and all discrepancies shall be appropriately documented via the query resolution process. Site monitors are appointed by the study sponsor and are independent of study site staff.

If electronic records are maintained, the method of verification must be determined in advance of starting the study.

At a minimum, source documents include the following information for each subject:

- Subject identification (name, sex, race)
- Documentation of subject eligibility
- Date of informed consent
- Dates of visits
- Documentation that protocol specific procedures were performed
- Results of study parameters, as required by the protocol
- IP accountability records
- Documentation of AEs and other safety parameters (if applicable)

- Records regarding medical histories and the use of concomitant therapies prior to and during the study
- Date of study completion and reason for early discontinuation, if applicable

It is required that the author of an entry in the source documents be identifiable. Direct access to source documentation (medical records) must be allowed for the purpose of verifying that the data recorded on the CRF are consistent with the original source data.

Only designated individuals at the site will complete the CRFs. The CRFs must be completed at regular intervals following the clinical study visit schedule. It is expected that all data reported have corresponding entries in the source documents. The principal investigator is responsible for reviewing and certifying that the CRFs are accurate and complete. The only subject identifiers recorded on the CRFs will be subject number, and subject demographic information.

#### 13.3 Data Review and Clarifications

A review of CRF data to the subject's source data will be completed by the site monitor to ensure completeness and accuracy. After the CRFs have been completed, additional data clarifications and/or additions may be needed as a result of the data cleaning process. Data clarifications are documented and are part of each subject's CRF.

# 13.4 Sponsor and Monitoring Responsibilities

The study sponsor will select principal investigators that are qualified by education, training, and experience to assume responsibility for the proper conduct of this clinical trial.

The study sponsor is financially funding this clinical trial and will compensate the investigator and/or the Institution(s) at which the study is conducted in accordance with a signed clinical trial agreement.

The study sponsor will designate a monitor to conduct the appropriate site visits at the appropriate intervals according to the study monitoring plan. The clinical investigation will be monitored to ensure that the rights and well-being of the subjects are protected, the reported data are accurate, complete, and verifiable from the source documents, and the study is conducted in compliance with the current approved protocol (and amendments[s], if applicable), with current GCP, and with applicable regulatory requirements.

The site may not screen subjects or perform the informed consent process on any subject until it receives a notification from an appropriate Study Sponsor representative that the site may

commence conducting study activities. Monitoring will be conducted periodically while the clinical study is ongoing. Monitoring methods may include site visits, telephone, written and fax correspondence. Close-out visits will take place after the last visit of the last subject at the site.

#### 13.5 Regulatory Documentation and Records Retention

The investigator is required to maintain up-to-date, complete regulatory documentation as indicated by the study sponsor and the investigator's files will be reviewed as part of the ongoing study monitoring. Financial information is to be kept separately.

Additionally, the investigator must keep study records and source documents consistent with the terms of the clinical study agreement with the study sponsor. If the investigator retires, relocates, or for any other reason withdraws from responsibility of keeping the study records, then the study sponsor must be notified and suitable arrangements made for retention of study records and source documents needed to comply with national and international regulations.

# 13.6 Quality Assurance and Quality Control

The study sponsor will secure agreement from all involved parties to ensure direct access to all study related sites, source data and documents, and reports for the purpose of monitoring and auditing by the study sponsor, and inspection by domestic and foreign regulatory authorities. Quality control will be applied to each stage of data handling to ensure that all data are reliable and have been processed correctly. Agreements made by the study sponsor with the investigator/institution and any other parties involved in the clinical study will be provided in writing as part of the protocol or as a separate agreement.

#### 14 ETHICS

Investigations are conducted in compliance with Good Clinical Practices; international and national regulations, laws, and guidelines; the conditions of approval imposed by reviewing IRBs/IECs or regulatory authorities; and in accordance with the ethical medical research principles outlined in the Declaration of Helsinki.

- The SOPs of the study sponsor and contract research organizations participating in the conduct of the clinical study and all other applicable regulations shall apply.
- Notifications and timelines for reporting protocol deviations should be based upon applicable Ethics Committee requirements.

The investigator must ensure that all personnel involved in the conduct of the study are qualified to perform their assigned responsibilities through relevant education, training, and

experience. The investigator and all clinical study staff must conduct the clinical study in compliance with the protocol. Deviations from this protocol, regulatory requirements, and/or GCP must be recorded and reported to the Sponsor prior to database lock. If needed, corrective and preventive action should be identified, implemented, and documented within the study records. Use of waivers to deviate from the clinical protocol is prohibited.

Before clinical study initiation, this protocol, the informed consent form, any other written information given to subjects, and any advertisements planned for subject recruitment must be approved by an IRB/IEC. The investigator must provide documentation of the IRB/IEC approval to the study sponsor. The approval must be dated and must identify the applicable protocol, amendments (if any), informed consent form, assent form (if any), all applicable recruiting materials, written information for subject, and subject compensation programs. The IRB/IEC must be provided with a copy of the IFU, any periodic safety updates, and all other information as required by local regulation and/or the IRB/IEC. At the end of the study, the investigator must notify the IRB/IEC about the study's completion. The IRB/IEC also must be notified if the study is terminated prematurely. Finally, the investigator must report to the IRB/IEC on the progress of the study at intervals stipulated by the IRB/IEC.

Voluntary informed consent must be obtained in writing from every subject. The obtaining of consent shall be documented before any procedure specific to the clinical investigation is applied to the subject.

The investigator must have a defined process for obtaining the required consent. Specifically, the investigator, or their delegate, must explain the clinical study to each potential subject and the subject must indicate voluntary consent by signing and dating the approved informed consent form. The subject must be provided an opportunity to ask questions of the investigator, and if required by local regulation, other qualified personnel. The investigator must provide the subject with a copy of the consent form written in a language the subject understands. The consent document must meet all applicable local laws and provide subjects with information regarding the purpose, procedures, requirements, and restrictions of the study, along with any known risks and potential benefits associated with the IP and the study, the available compensation, and the established provisions for maintaining confidentiality of personal, protected health information. Subjects will be told about the voluntary nature of participation in the study and must be provided with contact information for the appropriate individuals should questions or concerns arise during the study. The subject also must be told that their records may be accessed by appropriate authorities and sponsor-designated personnel. The investigator must keep the original, signed copy of the consent (file in

subject's medical records) and must provide a duplicate copy to each subject according to local regulations.

Human clinical trials liability insurance will be provided for participating subjects.

The study sponsor assures that the key design elements of this protocol will be registered on www.clinicaltrials.gov if required by current regulations and, if applicable, other public databases as required by local country regulations. In addition, results of this study will be made publicly available on www.clinicaltrials.gov regardless of outcome if required by current regulations and, if applicable, in other public databases as required by local country regulations.

#### 15 REFERENCES

#### 15.1 Regulations and Standards

The following references may be applicable in whole or in part for this clinical trial.

- ISO 11980:2012 Ophthalmic optics Contact lenses and contact lens care products -Guidance for clinical investigations
- EN ISO 14155:2020 clinical investigation of medical devices for human subjects Good Clinical Practice
- 21 CFR Part 11 Electronic Records; Electronic Signatures
- 21 CFR Part 50 Protection of Human Subjects
- 21 CFR Part 56 Institutional Review Boards
- 21 CFR Part 812 Investigational Device Exemptions
- 21 CFR Part 54 Financial Disclosure by Clinical investigators
- The California Bill of Rights, if applicable











